CLINICAL TRIAL: NCT03883724
Title: Impact of Behavioral Treatment of Insomnia on Nighttime Urine Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shachi Tyagi, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO18100572; R21AG060292 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-21 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Sleep Fragmentation; Poor Quality Sleep; Nocturia; Nocturnal Enuresis
Keywords: Nocturia; Poor sleep
MeSH Terms: conditions — Sleep Deprivation; Nocturia; Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief behavioral treatment for insomnia (Experimental): This group will undergo behavioral intervention proven to improve sleep among older adults: brief behavioral treatment for insomnia
  Interventions: Behavioral: Brief behavioral treatment of insomnia (BBTI)
- Information-only control (Other): This group is called information-only control. They will be provided sleep-related information. They will also view a video content of which overlap substantially with BBTI but without individualized behavioral instructions.
  Interventions: Behavioral: Information-only control (IC)

INTERVENTIONS:
Behavioral: Brief behavioral treatment of insomnia (BBTI) — The BBTI consists of a 45- to 60-minute individual intervention session followed by a 30-minute follow-up session 2 weeks later and 20-minute telephone calls after 1 and 3 weeks. The brief behavioral treatment component will focus on four behaviors that promote sleep through homeostatic, circadian, or association mechanisms. 50 These four interventions are simple to conceptualize and implement, and constitute the core of efficacious multi-modal behavioral treatments for insomnia.
  Arms: Brief behavioral treatment for insomnia
Behavioral: Information-only control (IC) — The IC condition is intended to emulate the behavioral treatment information generally to available patients. It includes instructions to review hand out on healthy sleep practices. We will also use patient education videos on insomnia developed locally and widely used in clinical research. The content of these videos overlap substantially with BBTI but without individualized behavioral instructions. Two weeks later, IC participants will receive a 10-minute follow-up telephone call to encourage continued participation. Participants will be referred to the brochures for specific sleep-related questions.
  Arms: Information-only control

SUMMARY:
Nocturia is prevalent in older adults and it vastly reduces quality of life. Yet its treatment remains inadequate because its causes are not well understood, especially nocturnal polyuria or increased urine production at night. This study, which builds on the investigators' ongoing research, would be the first of its kind to explore the role of sleep in nighttime urine production. The findings will contribute important knowledge to guide development of better targeted and more effective therapy for this prevalent and morbid condition.

DETAILED DESCRIPTION:
Prevalent, morbid, and costly ($61 billion/year in 2012), nocturia is a major problem, especially for older adults. It increases the risk of falls, fractures, depression, nursing home placement, and death. Yet management of nocturia remains inadequate. Most behavior and pharmacotherapies for nocturia focus on bladder-related etiologies, and it's most prevalent attribute nocturnal polyuria (NP), or increased urine production during sleep remains poorly understood and inadequately treated with little advancement over the last 50 years. Disruption of diurnal excretory pattern, with higher nighttime urine production is common in older adults. While studies in young adults show that sleep plays a critical role in regulating nighttime urine production, among older adults the role of poor sleep in NP is under-investigated.

Urine production follows a circadian pattern in which transition from wake to sleep is followed by a pronounced decrease in excretion of water, electrolytes and other osmotically active substances. Studies in young population have established that physiological urine production follows a circadian rhythm, which is regulated by diurnal variation in secretion of hormones controlling water and salt excretion such as arginine vasopressin, renin-angiotensin-aldosterone system, and atrial natriuretic peptide. Sleep deprivation blunts nocturnal surge of these hormones and consequently alter water and salt excretion thereby increase nighttime urine volume leading to NP.

Recent evidence suggests that poor sleep quality, frequent sleep interruptions especially in the first part of the night and shorter duration of first uninterrupted sleep period are associated with NP but its pathophysiology is not fully understood. Additionally, among older adults with poor sleep, the investigators have shown that a behavioral intervention directed solely towards sleep (BBTI- brief behavioral treatment of insomnia an efficacious multimodal behavioral treatment for insomnia) not only improves sleep, but also nocturia. Hence, the investigators postulate that sleep interruptions in the first part of the sleep impacts the hormonal regulation of nighttime urine production causing NP. In addition, the investigators postulate that interventions to prolong the first uninterrupted sleep period will decrease NP and hence nocturia.

The, aims of the present proposal are to: 1) examine the impact of BBTI on duration of the first of uninterrupted sleep period and NP in elderly with nocturia; and 2) establish NP and duration of first uninterrupted sleep as mechanisms by which BBTI impacts nocturia. The investigators' hypothesis is that BBTI improves nocturia not only by improving sleep, (and specifically, duration of the first uninterrupted sleep period), but also by decreasing NP.

To accomplish these goals the investigators will recruit 60 community dwelling adults (aged >65) with nocturia and NP. Sleep will be assessed subjectively with the Insomnia Severity Index and objectively by 7-day sleep diary and wrist actigraph. Concurrently the investigators will collect 3-day bladder diary data to document their voiding pattern and volume during day and night. Participants will be randomized to receive the 4-week behavioral sleep intervention BBTI by a trained therapist or an information control intervention. The participants will repeat the study measures post-intervention.

The study results will provide important insights into shared pathological mechanisms underlying poor sleep, nocturia and nighttime urine production.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory and functionally-independent community-dwelling men and women
* aged 65 years, or more
* with nocturia ≥2/night
* poor sleep because of frequent awakenings

Exclusion Criteria:

* Unstable or acute medical or central nervous system conditions
* Untreated, current, severe psychiatric condition
* Untreated, current, severe overactive bladder syndrome
* Post void residual > 30ml
* Sleep apnea with AHI≥15
* Currently diagnosed and/or treated Obstructive Sleep Apnea, Restless Legs Syndrome, parasomnia
* Congestive heart failure, by exam or Beta natriuretic peptide (BNP)> 30 pmol/L
* Chronic kidney disease, stage III-V (eGFR<50)
* >14 alcohol drinks per week

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shachi Tyagi, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started Jan 2019 through April 2021. The initial screening was completed telephonically and once screened eligible, the interested participants underwent study related assessments and procedures at the study research suite - Continence Research Unit at UPMC Montefore Hospital located in Pittsburgh, PA
Pre-assignment Details: After the telephone screening, the eligible participants completed a home sleep apnea assessment using device ApneaLink Air that was sent to them via mail with instructions for use at home. Those with AHI≥15 were excluded per study exclusion criteria before the in-person Visit 1 or signing the informed consent.
Period: Overall Study
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall, 56 participants were eligible, 29 randomized to BBTI and 27 to control group
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 29 | 27 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 27.2 (5.7) | 28.4 (5.1) | 27.8 (5.4)
Post void residual [Mean (Standard Deviation); unit: ml] | 11.6 (18.5) | 19.3 (28.8) | 15.2 (24)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.86 (0.21) | 0.94 (0.23) | 0.9 (0.2)
Calcium channel blocker [Count of Participants; unit: Participants] | 3 | 4 | 7
Beta-blocker [Count of Participants; unit: Participants] | 2 | 7 | 9
ACE-I/ARB [Count of Participants; unit: Participants] | 7 | 5 | 12
Thiazide diuretic [Count of Participants; unit: Participants] | 4 | 5 | 9
Loop diuretic [Count of Participants; unit: Participants] | 2 | 2 | 4
Anti-depressant [Count of Participants; unit: Participants] | 3 | 4 | 7
NSAIDS [Count of Participants; unit: Participants] | 6 | 4 | 10
Proton pump inhibitor/ H2 blocker [Count of Participants; unit: Participants] | 6 | 5 | 11
Antimuscarinic [Count of Participants; unit: Participants] | 1 | 1 | 2
Alpha-blocker [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Nocturnal Polyuria Index
Description: Nocturnal Polyuria Index (NPI) is the percentage of 24-hour urine production excreted at night. It is measured using 3-day bladder diary that participants will complete pre- and post-intervention in which the participants document the time and volume of each void during the day and night for 3 days. NPI is calculated using a) nocturnal urine volume (determined by adding the volume of all voids between the times marked in the bladder diary as going to bed with the intent of sleeping and the first awakening to void. The first void after waking is included in the nighttime urine volume), and b) 24-hour urine volume. NPI is calculated as: nocturnal urine volume /24-hour urine volume
Time Frame: change from baseline nocturnal polyuria index at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of urine volume
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control
Number analyzed (Participants) | 29 | 27
percentage of urine volume
  Pre-intervention | 41.7 (9.9) | 41.7 (10.1)
  Post-intervention | 34.5 (13) | 37.8 (8.6)
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia vs Information-only Control; Change in NPi pre- vs post-intervention comparing between group analysis; Test type: Other — ANCOVA between-group analysis was completed comparing of Pre- to Post-Intervention change adjusting for baseline value of the outcome; p = 0.3, ANCOVA; between-group analysis was completed comparing of Pre- to Post-Intervention change adjusting for baseline value of the outcome

2. Secondary Outcome: Change in Nocturia
Description: Nocturia=number of awakenings to void each night
Time Frame: change from baseline nocturia episodes each night at 4 weeks
Measure: Mean (Standard Deviation); unit: awakenings, as reported on bladder diary
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control
Number analyzed (Participants) | 29 | 27
awakenings, as reported on bladder diary
  Pre-intervention | 2.3 (.6) | 2.1 (.7)
  Post-intervention | 1.3 (.6) | 1.8 (.6)
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia vs Information-only Control; Change in nocturia frequency pre- vs post-intervention comparing between group analysis; Test type: Other — [test comment as in outcome 1, analysis 1]; p < .01, ANCOVA — Change in nocturia frequency pre- vs post-intervention comparing between groups BBTI vs IC; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Duration of Uninterrupted Sleep
Description: Duration of uninterrupted sleep is the first uninterrupted sleep period before first awakening to void
Time Frame: Change from baseline duration of uninterrupted sleep at 4 weeks
Measure: Mean (Standard Deviation); unit: minutes, imputed from bladder diary
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control
Number analyzed (Participants) | 29 | 27
minutes, imputed from bladder diary
  Pre-intervention | 174 (53) | 188 (53)
  Post-intervention | 227 (68) | 210 (72)
Statistical Analysis 1: Comparison: Brief Behavioral Treatment for Insomnia vs Information-only Control; between-group analysis was completed comparing of Pre- to Post-Intervention change adjusting for baseline value of the outcome; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.3, ANCOVA; ANCOVA between-group analysis was completed comparing of Pre- to Post-Intervention change adjusting for baseline value of the outcome

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of study participation for each participant, 6-8 weeks
Description: Adverse events were noted by self-report from participants. Specific worsening of any sleep related issues were specifically asked during the telephonic follow-up every 2 visits following randomization.
Arm/Group | Brief Behavioral Treatment for Insomnia | Information-only Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT03883724/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03883724/ICF_001.pdf